CLINICAL TRIAL: NCT04865887
Title: A Phase II Trial of Combination Therapy of Pembrolizumab and Lenvatinib in Patients With Locally Advanced or Metastatic Cervical Cancer
Brief Title: Pembrolizumab and Lenvatinib in Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003849; MK-3475-A70 (Other: Funding source)
Record Dates: First submitted 2021-04-16; First posted 2021-04-29 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cervical Cancer; Metastatic Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab with Lenvatinib (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — 200mg, every 3 weeks, IV infusion
Drug: Lenvatinib — 20 mg (2 capsules x10mg), daily, orally

SUMMARY:
This is a phase II trial of combination therapy of pembrolizumab and lenvatinib in patients with locally advanced or metastatic cervical cancer that had failed first line of therapy. The hypothesis is the combination of lenvatinib and pembrolizumab will overcome vascular endothelial growth factor (VEGF)-mediated immunosuppression to enhance the response of patients with locally advanced or metastatic cervical cancer.

DETAILED DESCRIPTION:
The primary endpoint of this phase II study is to determine the objective response rate (partial response [PR] + complete response [CR]) of specific pembrolizumab-lenvatinib combination therapy in patients with locally advanced or metastatic cervical cancer. The phase II portion of the trial will follow Simon's minimax two-stage design1.

In the Stage 1, 11 patients will be accrued. If 1 or fewer patients among these 11 patients achieve an objective response with the pembrolizumab-lenvatinib combination therapy, the combination therapy will be rejected and the trial stopped. However, if there are 2 or more patients who exhibit response in the Stage 1, then an additional 24 patients will be entered into the Stage 2, for a total of 35 patients in this phase II study. If 9 or more patients exhibit response among these 35 patients, then the treatment will be considered for further investigation. Any unplanned interim analysis will utilize the sequential conditional probability ratio test (SCPRT)2, which allows an early assessment of statistical evidence for both efficacy and futility, and provides a discordance probability that early trend could be reversed should the trial continue to enroll all 35 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of locally advanced or metastatic cervical cancer will be enrolled in this study.
2. Patients with progression or intolerance to at least one line of therapy in the locally advanced or metastatic setting will be eligible for this study.
3. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined OR
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
5. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue. Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 28 days prior to the date of treatment initiation.
8. Have adequate organ function as defined. Specimens must be collected within 28 days prior to the start of study treatment.

   1. Absolute neutrophil count (ANC) ≥1500/µL
   2. Platelets ≥100 000/µL
   3. Hemoglobin ≥9.0 g/dL
   4. Creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
   5. Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
   6. AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
   7. International normalized ratio (INR) OR prothrombin time (PT), Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment initiation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent.
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
5. Has received a live vaccine or live attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma) that have undergone potentially curative therapy are not excluded.
9. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab or lenvatinib and/or any of their excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV).
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
19. Has uncontrolled blood pressure (BP) (Systolic BP>140 mmHg or diastolic BP>90 mmHg) in spite of an optimized regimen of antihypertensive medication.
20. Has electrolyte abnormalities that have not been corrected.
21. Has significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening.
22. Has bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
23. Subjects having > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
24. Has gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
25. Prolongation of QTc interval to >480 ms.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 2 years
  To evaluate the clinical activity (as assessed by objective response rate [ORR]) of specific pembrolizumab-lenvatinib combination.

SECONDARY OUTCOMES:
Duration of response | up to 2 years
  To evaluate the clinical activity (as assessed by duration of response (DoR)) of pembrolizumab-lenvatinib combinations. DOR: length of time tumor continues to respond to the treatment.
Progression Free survival | up to 2 years
  To evaluate the clinical activity (as assessed by progression-free survival [PFS]) of pembrolizumab-lenvatinib combinations. PFS: Time from treatment initiation to the first documented disease progression per response evaluation criteria in solid tumors (RECIST) 1.1 as assessed by local site or death, whichever occurs first.
Overall survival | Cycle 1 Day 1, Day 1 of each cycle (each cycle is 21 days), every 12 weeks after end of treatment
  To evaluate the clinical activity (as assessed by overall survival [OS]) of pembrolizumab-lenvatinib combinations. OS: Time from treatment initiation to death due to any cause.
Incidence of adverse events | Day 1 of each cycle (each cycle is 21 days), up to 2 years
  To evaluate the safety and tolerability of pembrolizumab-lenvatinib combination:
  Number of Participants Experiencing Adverse Events (AEs) according to NCI CTCAE Version 5.0.
Incidence of study drug discontinuation due to Adverse Events | Day 1 of each cycle (each cycle is 21 days), up to 2 years
  To evaluate the safety and tolerability of pembrolizumab-lenvatinib combination: Number of Participants Discontinuing Study Drug Due to AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Khleif, MD, Principal Investigator — Georgetown University
Locations (4):
- United States (4):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No